CLINICAL TRIAL: NCT06669260
Title: Prospective Study to Evaluate QoL Scores and Post-operative Complications Using TEThA (Transfixing Endovenous Thermal Ablation) Technique in Tributary Veins Treatment
Brief Title: Evaluating QoL and Postoperative Complications Using TEThA Technique in the Treatment of Tributary Veins
Acronym: TEThA
Status: Not yet recruiting | Type: Observational
Sponsor: Nara Medeiros Cunha de Melo Vasconcelos (Other)
Collaborators: Gabriela de Oliveira Buril (Unknown); Marcelo Halfen Grill (Unknown)
Responsible Party: Sponsor-Investigator, Nara Medeiros Cunha de Melo Vasconcelos, MD, Science Valley Research Institute
Organization: Science Valley Research Institute (Other)
Other Study IDs: TEThA
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Varicose Veins; Quality of Life; Laser
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TEThA technique: TEThA technique
  Interventions: Procedure: TEThA technique

INTERVENTIONS:
Procedure: TEThA technique — Patient in an orthostatic position, previously marked varicose veins will be punctured with a tracing adjacent to them, surrounding their edges. Applying an augmented reality device and Doppler ultrasound (Doppler USG), the marking will be complemented in the supine position. These punctures will in turn be carried out using the TEThA technique - endovenous thermoablation of tributary veins by means of transfixation - and will be done sequentially as they are treated one by one with endo- and perivenous thermoablation under generous tumescence with 0.08% lidocaine in saline solution. The laser used to treat the tributary veins will also be 1470 nm and will be fired as the fiber is removed at a speed of 1 mm/sec and power ranging from 5 to 7 watts.

SUMMARY:
Endovenous laser thermoablation is a well-established alternative for the treatment of tributary veins. We believe that it is possible to improve the techniques described in the literature, aiming not only to allocate the laser fiber within the venous lumen, but mainly to transfix the vessel walls - a technique called TEThA (Transfixing Endovenous Thermal Ablation).

DETAILED DESCRIPTION:
Endovenous laser thermoablation is an alternative for the treatment of tributary veins that is not yet one of the main alternatives in our specialty's consensus. In order to treat tributary veins applying laser, several punctures and the complete placement of introducer catheters are recommended in order to position the endolaser fiber in the lumen of the varicose vein before performing thermoablation of the saphenous veins. However, we believe that it is possible to perform an adequate treatment with a smaller number of punctures, aiming not only to place the laser fiber inside the venous lumen, but mainly to transfix the vessel walls - a technique called TEThA (Transfixing Endovenous Thermal Ablation). Our aim is to carry out a prospective cohort study to assess the Aberdeen score in patients undergoing the TEThA technique for the treatment of tributary veins.

ELIGIBILITY:
Inclusion Criteria:

Patients with varicose veins > 2mm associated with reflux of great or small saphenous veins with CEAP C2 to C6

Exclusion Criteria:

Patients under 18 years Acute or previous thrombophlebitis or deep vein thrombosis. Pregnant patient. Reject the Informed Consent Form.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with tributary veins bigger than 2mm, presenting saphenous truncal incompetency scoring from C2 to C6 in CEAP
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-21 (Estimated); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Quality of Life score using Aberdeen Varicose Veins Questionnaire (AVVQ) | Baseline, Timepoints post-procedire: 1 month, 3 months, 6 months
  AVVQ is an easy-to-administer, self-administered instrument, it consists of 3 dimensions, which are physical, sociofunctional and psychological. It is interpreted through a score, which can vary between 0 and 100, with 0 representing no evidence of varicose veins and 100 the most serious problem associated with varicose veins.
Quality of life score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) | Timepoints post-procedire: 1 month, 3 months, 6 months
  CIVIQ-14 is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe). Based on inputs, Global Index Score (GIS) will be tabulated, ranging from 0 to 100 - the higher the value, the poorer the quality of life.

SECONDARY OUTCOMES:
Hyperpigmentation | Baseline, 30 days and 180 days
  Presence or absence of hyperpigmentation in the limb treated by a endovenous laser with TEThA tecnique (phototodocumentation, US Doppler)
Presence of induration | 30 days and 180 days
  Induration noticed on the saphenous vein path (phototodocumentation, US Doppler)
Presence of Paresthesia | 30 days and 180 days
  Presence or absence of paresthesia in the limb treated by endovenous laser TEThA technique
Skin burns | 7 days
  Presence or absence of skin burns in the limb treated by a endovenous laser with TEThA technique
Lymphedema | 30 days and 180 days
  Presence or absence of lymphedema diagnosed by exam of lymphoscintigraphy in the limb treated by endovenous laser TEThA technique
Sclerothrombus | 7 days
  Presence of Sclerothrombus (US doppler)
Complementary treatment | 180 days
  Percentage of participants with residual veins

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salim S, Machin M, Patterson BO, Onida S, Davies AH. Global Epidemiology of Chronic Venous Disease: A Systematic Review With Pooled Prevalence Analysis. Ann Surg. 2021 Dec 1;274(6):971-976. doi: 10.1097/SLA.0000000000004631. PMID 33214466
- [Background] Lurie F, Passman M, Meisner M, Dalsing M, Masuda E, Welch H, Bush RL, Blebea J, Carpentier PH, De Maeseneer M, Gasparis A, Labropoulos N, Marston WA, Rafetto J, Santiago F, Shortell C, Uhl JF, Urbanek T, van Rij A, Eklof B, Gloviczki P, Kistner R, Lawrence P, Moneta G, Padberg F, Perrin M, Wakefield T. The 2020 update of the CEAP classification system and reporting standards. J Vasc Surg Venous Lymphat Disord. 2020 May;8(3):342-352. doi: 10.1016/j.jvsv.2019.12.075. Epub 2020 Feb 27. PMID 32113854
- [Background] De Maeseneer MG, Kakkos SK, Aherne T, Baekgaard N, Black S, Blomgren L, Giannoukas A, Gohel M, de Graaf R, Hamel-Desnos C, Jawien A, Jaworucka-Kaczorowska A, Lattimer CR, Mosti G, Noppeney T, van Rijn MJ, Stansby G, Esvs Guidelines Committee, Kolh P, Bastos Goncalves F, Chakfe N, Coscas R, de Borst GJ, Dias NV, Hinchliffe RJ, Koncar IB, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, Bjorck M, Labropoulos N, Lurie F, Mansilha A, Nyamekye IK, Ramirez Ortega M, Ulloa JH, Urbanek T, van Rij AM, Vuylsteke ME. Editor's Choice - European Society for Vascular Surgery (ESVS) 2022 Clinical Practice Guidelines on the Management of Chronic Venous Disease of the Lower Limbs. Eur J Vasc Endovasc Surg. 2022 Feb;63(2):184-267. doi: 10.1016/j.ejvs.2021.12.024. Epub 2022 Jan 11. No abstract available. PMID 35027279
- [Background] Vasconcelos NMCM, Kumakura HS, Grill MH, Silva MCE. Treatment of the small saphenous vein and tributary veins with endolaser associated with ultrasound-guided foam in a patient with post-thrombotic syndrome: presenting the TEThA technique. J Vasc Bras. 2024 Nov 29;23:e20230142. doi: 10.1590/1677-5449.202301422. eCollection 2024. PMID 39629276